CLINICAL TRIAL: NCT03764124
Title: Prospective Monocentric Observational Study of Kidney Transplant Recipients at the CHU of Liege for the Prediction of Allograft Survival and Impact of Imaging in Clinical Decision-making.
Brief Title: Observation Study for Prediction of Allograft Survival and Impact of Imaging in Kidney Transplant Recipients.
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Antoine Bouquegneau, MD, University of Liege
Other Study IDs: Liège KO
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplantation
Keywords: Allograft survival; PET/CT imaging; Corticoids withdrawal; Bone mineral Density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney recipients: Kidney recipients aged over 18 and of all sexes recruited between 2007 and 2020 from the Centre Hospitalier Universitaire de Liege, who have e-GFR follow-up and data from protocol and for cause biopsies available at 1-year post transplant. PET/CT imaging will be performed with patient's approval for protocol and per cause biopsies we performed. Data will be collected in the follow up such as clinical, biological and histological data.
  Interventions: Diagnostic Test: PET/CT imaging

INTERVENTIONS:
Diagnostic Test: PET/CT imaging — The PET/CT procedure was performed using cross-calibrated Philips Gemini TF Big Bore or TF 16 PET/CT systems (Philips Medical Systems, Cleveland, OH) at 201 18 minutes following intravenous injection of a mean dose of 3.2 0.2 MBq/kg of body weight of 18 F-FDG. A low-dose helical CT (5-mm slice thickness, 120-kV tube voltage, and 40-mAs tube current-time product) centered to the renal transplant was performed, followed by PET scanning with two bed positions, each lasting 240 seconds. Images were reconstructed using iterative list mode time-of-flight algorithms. Corrections for attenuation, dead time and random and scatter events were applied.

SUMMARY:
To further develop personalized medicine in kidney transplantation and improve transplant patient outcomes, attention has been given to define early surrogate endpoints that might aid therapeutic interventions, and help clinical decision-making.

To adequately predict transplant patients' individual risks of allograft loss and patients' complications, this would require a complex integration of data, including: donor data, recipient characteristics, transplant characteristics, biopsies results, immunosuppressive regimen, allograft infections, acute kidney injuries, recipient immune profiles, protocol and per cause biopsies and imaging (PET/CT imaging).

This project aims:

1. Assessed the usefulness of 18F-FDG PET/CT imaging in kidney transplantation recipients presenting with suspected acute rejection who underwent a transplant needle biopsy;
2. To develop a prognostic risk score to predict kidney allograft survival;
3. To evaluate the impact of corticoids withdrawal on long term outcomes (risk of rejection and impact on bone mineral density);
4. Evaluate the type and the frequencies of complications in our kidney transplant population

DETAILED DESCRIPTION:
1. The detection of acute rejection in kidney transplant recipients, depends critically on assessments of serum creatinine, an insensitive measure of renal injury and the diagnosis relies on renal transplant needle biopsy which is an invasive procedure associated with a significant risk of bleeding and graft loss and is limited by sampling error and/or interobserver variability. Moreover, repeated biopsies to evaluate a renal graft's status pose challenges, including practicability and cost. Consequently, other sensitive and less invasive modalities, including gene expression profiling and omic analyses of blood and urine samples as well as in vivo imaging, are currently under investigation to reinforce our clinical armamentarium for acute rejection diagnosis. Likewise, it would be useful to non-invasively predict rejection in kidney transplant recipients with acute renal dysfunction and suspected acute rejection, thereby avoiding unnecessary transplant biopsy.
2. This study aims to generate a scoring system that predicts individual patients' risk of long-term kidney allograft failure.
3. Since 2007, the protocol in our institution is to withdraw the corticoids after 3 months after the protocol biopsy if no sign of rejection is demonstrated. We would like to evaluate the impact of such decision in the risk of rejection and the long-term allograft outcome in our patients. We are looking also to the impact on bone mineral density after corticoids withdrawal in those patients.
4. Evaluate the type and the frequencies of complications in our kidney transplant population to adapt our daily basis clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipient transplanted after 2007
* Kidney recipient over 18 years of age
* Clinical, biological, immunological and follow up data available

Exclusion Criteria:

* Combined transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney recipients aged over 18 of all sexes recruited between 2007 and 2020 from the Centre Hospitalier Universitaire of Liege, who have e-GFR follow-up and data from protocol and for cause biopsies available at 1-year post transplant. PET/CT imaging will be performed with patient's approval for protocol and per cause biopsies we performed. Data will be collected in the follow up such as clinical, biological and histological data.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Imaging | Prediction of rejection at time of biopsies
  Prediction model of the PET/CT imaging to predict the histological results of a biopsy.

SECONDARY OUTCOMES:
Allograft survival probability post transplantation | Allograft survival probability at 1-year post transplantation
  Allograft survival probability calculated from clinical, histological, immunological, and functional variables assessed at the time of transplant and at the time of biopsy at 3-months post transplant.
Rejection | Evaluation of the risk of rejection during follow-up in patients with corticoids withdrawal at 3 months post transplantation
  Risk of rejection rate in patients with corticosteroids withdrawal at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS JOURET, PhD, Principal Investigator — CHU Liege department of Nephrology-Dialysis and Transplantation, and Groupe Interdisciplinaire de Géno-protéomique Appliquée, Cardiovascular Sciences.
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No